CLINICAL TRIAL: NCT03989973
Title: West China Hospital, Sichuan University
Brief Title: Two-dimensional Shear-Wave Elastography Evaluate Esophageal Varices Bleeding Risk of Liver Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, luo xuefeng, Associate Professor, West China Hospital
Other Study IDs: 2D-SWE evaluate varices
Record Dates: First submitted 2019-06-16; First posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Liver Cirrhosis; Esophageal Varices; Liver Stiffness
Keywords: Liver cirrhosis; Esophageal Varices; Liver Stiffness; Spleen Stiffness
MeSH Terms: conditions — Liver Cirrhosis; Esophageal and Gastric Varices | interventions — Gastroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cirrhosis patients: Patients were diagnosed by liver biopsy, CT or ultrasound
  Interventions: Diagnostic Test: Gastroscopy

INTERVENTIONS:
Diagnostic Test: Gastroscopy — Gastroscopy

SUMMARY:
The purpose of this retrospective study was to investigate the diagnostic performance of 2D-SWE for predicting the presence of esophageal varices and high-risk varices in patients with liver cirrhosis.

DETAILED DESCRIPTION:
Variceal bleeding is a fatal complication in patients with liver cirrhosis. A screening esophagogastroduodenoscopy (EGD) is recommended in all patients with cirrhosis to identify those patients at risk of variceal bleeding. However, this technique is invasive, uncomfortable and costly. Moreover, with the development of noninvasive technology for early diagnosis of liver cirrhosis, half of these patients will not develop varices within 10 years and therefore will undergo unnecessary EGD screening. Thus, the need for noninvasive screening methods for varices in patients with cirrhosis is urgent.

2D-SWE is a promising new type of shear wave-based ultrasound technique for measuring LS. The shear waves are generated directly within the tissue by acoustic radiation force impulse, allowing the measurement of stiffness in patients with ascites. In addition, the LS values can be obtained on the basis of anatomic information to avoid major vessels and control major measurement bias. 2D-SWE has been reported to have high reliability and reproducibility in assessing liver stiffness. Several studies compared TE with 2D-SWE in predicting fibrosis stages and portal hypertension, which suggested that 2D-SWE has a higher technical success rate and a better diagnostic value for portal hypertension than TE.The purpose of this retrospective study was to investigate the diagnostic performance of 2D-SWE for predicting the presence of esophageal varices and high-risk varices in patients with liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis were diagnosed by liver biopsy, CT and ultrasound before enrolled
* Age was 16-80

Exclusion Criteria:

* With bleeding history
* With EVL history, BRTO or TIPS history
* With NSBB history
* With ascites
* With splenectomy or splenic embolism, history
* With liver cancer

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: compensated cirrhosis
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Liver Stiffness | 1 day (At 2D-SWE scanning time)
  Liver stiffness assessed by 2D-SWE
Varices stage | 1 day (At gastroscopy performed time)
  Gastroscopy was used to assess varices stage

CONTACTS AND LOCATIONS:
Overall Officials: Xuefeng Luo, Principal Investigator — West China Hospital of Sicuan Univerisity
Locations (1):
- West China Hospital of Sichuan Univerisity, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No